CLINICAL TRIAL: NCT05816070
Title: A Phase II, Multi-Center, Randomized, Parallel Controlled Study to Evaluate the Clinical Efficacy and Safety of IVIEW 1201 Compared to Ofloxacin Eye Drops in the Treatment of Acute Bacterial Conjunctivitis
Brief Title: Trial to Evaluate the Efficacy and Safety of IVIEW-1201 in Acute Bacterial Conjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IVIEW Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IVIEW-1201-BAC-II
Record Dates: First submitted 2023-03-29; First posted 2023-04-18 (Actual); Results first posted 2025-06-15 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Acute Bacterial Conjunctivitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IVIEW-1201 (Experimental)
  Interventions: Drug: IVIEW-1201
- Ofloxacin Eye Drops (Active Comparator)
  Interventions: Drug: Ofloxacin Eye Drops

INTERVENTIONS:
Drug: IVIEW-1201 — Four times per day for day 1-2 and three times per day for day 3-7
  Arms: IVIEW-1201
Drug: Ofloxacin Eye Drops — Four times per day for day 1-2 and three times per day for day 3-7
  Arms: Ofloxacin Eye Drops

SUMMARY:
A Phase 2, Multi-center, Randomized, Parallel Controlled Study to Evaluate the Clinical Efficacy and Safety of IVIEW-1201 (1.0% Povidone-Iodine) Gel Forming Ophthalmic Solution Compared to Ofloxacin Eye Drops in the Treatment of Acute Bacterial Conjunctivitis

ELIGIBILITY:
Inclusion Criteria:

1. Volunteered to participate in the study and signed the Informed Consent Form after receiving a verbal and written explanation of this clinical trial. In cases where the subject is unable to sign the Informed Consent Form, his/her guardian may sign in accordance with relevant regulations.
2. Aged above 15 ( inclusive), male or female.
3. A diagnosis of acute bacterial conjunctivitis based on clinical observations:

   1. a score of ≥1 for bulbar conjunctival congestion and ≥1 for conjunctival secretion/exudation in at least one eye (same eye);
   2. increased purulent, mucopurulent or mucopurulent secretions are observed in the conjunctival sac of the affected eye in all patients.
4. Willing to cooperate in the completion of all procedures and visits required for the trial.

Exclusion Criteria:

1. Patients with systemic or ocular diseases, or functional disorders with comorbidities, or structural abnormalities that, in the judgment of the investigator, could adversely affect the course or results of the trial (e.g., hyperthyroidism, hepatitis, acute and chronic renal insufficiency).
2. Those who have a history of allergy or serious adverse reactions to any component of IVIEW 1201 (1.0% povidone iodine ophthalmic gel sterile solution) and Of laxacin Eye Drops; have a history of allergy or serious adverse reactions to quinolones; or have a cumulative total of three or more allergies to other drugs, food and environment; or who are prone to allergic symptoms such as rash and urticaria;
3. Symptoms or signs of bacterial conjunctivitis for more than 72 hours prior to screening;
4. Suspected fungal, viral or acanthamoeba infections based on clinical observations;
5. Those with severe keratitis or corneal opacity affecting the study results;
6. Active inflammation of the cornea, iris, or anterior chamber;
7. Corrected visual acuity of less than 0.2 in either eye;
8. History of eye surgery within 3 months prior to screening;
9. Those who have a history of acute or chronic dacryocystitis;
10. Those who need to wear corneal contact lenses during the trial;
11. Those who have used antibiotic eye drops or glucocorticoid eye drops within 14 days, and oral or intravenous antibiotics within 72 hours prior to screening;
12. Systemic use of steroidal drugs within 14 days prior to screening. Local use of eye steroidal drugs or nonsteroidal anti-inflammatory drugs (NSAIDs) within 7 days before enrollment (nasally or bronchially inhaled steroidal drugs are not allowed during the study);
13. Those with co-infections requiring treatment with other anti-infective drugs in the study;
14. Those who are using other drugs that may interfere with the efficacy or safety evaluation of the drug;
15. Participation in other interventional clinical trials within 30 days prior to the study;
16. Pregnant or lactating women, women with positive pregnancy tests and those planning to become pregnant (including male subjects); subjects who do not take effective contraceptive measures within 1 month before enrollment, or subjects (including male subjects) who are unwilling to take effective contraceptive measures within the next 6 months.
17. Other conditions or illnesses judged by the clinical investigator to be unsuitable for enrollment.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2024-10-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital of Shandong First Medical University, Jinan, Shandong, China

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All sites recruited participants simultaneously. They might have the same/ very close enrollment dates. So the final enrollments (129 participants) exceeded the proposed number (120 participatns in protocol) because a couple of participants were enrolled at similar time when approaching to the end of enrollment.
Period: Overall Study
Arm/Group | IVIEW-1201 | Ofloxacin Eye Drops
Started | 65 | 64
Completed | 63 | 62
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- IVIEW-1201; Ofloxacin Eye Drops: Administed once at the study site, and then at least 3 hours apart until bedtime, with a maximum of 4 doses on D1; 4 times on D2 at least 3 hours apart; 3 times a day at least 3 hours apart from D3 to D7. The duration of treatment is 7 days.
- Total: Total of all reporting groups
Arm/Group | IVIEW-1201 | Ofloxacin Eye Drops | Total
Number analyzed (Participants) | 65 | 64 | 129
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.60 (14.58) | 56.06 (13.83) | 56.84 (14.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 36 | 77
  Male | 24 | 28 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Han | 61 | 62 | 123
  Ethnicity: Others | 4 | 2 | 6
Height [Mean (Standard Deviation); unit: cm] | 163.43 (7.52) | 165.13 (8.10) | 164.27 (7.83)
Weight [Mean (Standard Deviation); unit: kg] | 64.69 (11.07) | 64.68 (11.10) | 64.68 (11.04)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure Rate
Description: The proportion of subjects with a score of 0 (0=Absent, 1=Mild, 2=Moderate, 3=Severe.) for bulbar conjunctival congestion and 0 (0=Absent, 1=Mild, 2=Moderate, 3=Severe.) for conjunctival secretion/exudation at Visit 4 (Day 8±1), Visit 5 (Day 14±1).
Time Frame: Take the visit 4 (Day 8±1) data, unless the subject was not cured and did not continue the treatment after visit 4 (Day 8±1) , in which case, visit 5 (Day 14±1) data would be used instead of Visit 4 data (Day 8±1).
Measure: Count of Participants; unit: Participants
Arm/Group | IVIEW-1201 | Ofloxacin Eye Drops
Number analyzed (Participants) | 64 | 64
Participants
  Clinically Cured | 37 | 31
  Not Clinically Cured | 27 | 33
Statistical Analysis 1: Comparison: IVIEW-1201 vs Ofloxacin Eye Drops; Test type: Non-Inferiority — The non-inferiority margin is -10% based on the general standard of antibacterial drug. Non-inferiority is established when P<0.05; p = 0.0137, Chi-squared

2. Secondary Outcome: Clearance Rate
Description: Bacterial clearance is defined as positive bacterial culture at baseline and negative bacterial culture at the last visit.
Time Frame: Day 3, Day 6, Day 8±1, Day 14±1
Measure: Count of Participants; unit: Participants
Arm/Group | IVIEW-1201 | Ofloxacin Eye Drops
Number analyzed (Participants) | 42 | 42
Participants
  Day 3: Cleared | 23 | 33
  Day 3: Not Cleared | 19 | 9
  Day 6: Cleared | 21 | 33
  Day 6: Not Cleared | 21 | 9
  Day 8±1: Cleared | 25 | 37
  Day 8±1: Not Cleared | 17 | 5
  Day 14±1: Cleared | 30 | 34
  Day 14±1: Not Cleared | 12 | 8

ADVERSE EVENTS:
Time Frame: Through participants completion of the study, an average of 2 weeks.
Arm/Group | IVIEW-1201 | Ofloxacin Eye Drops
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/64
Serious Adverse Events (participants affected / at risk) | 1/64 | 0/64
Other Adverse Events (participants affected / at risk) | 11/64 | 0/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVIEW-1201 (N=64) | Ofloxacin Eye Drops (N=64)
Pneumonia infection (Infections and infestations) | 1 (1) | 0 (0) — The subject was diagnosed with pneumonia [a Grade 3 AE leading to hospitalization (outcome: resolved), but not related to the investigational drug] and did not withdraw from the trial due to the SAE.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVIEW-1201 (N=64) | Ofloxacin Eye Drops (N=64)
Eye Pain (Eye disorders) | 11 (11) | 0 (0) — In the study, all the AEs with an incidence ≥ 5% were eye pain and occurred in the treatment group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT05816070/Prot_SAP_000.pdf